CLINICAL TRIAL: NCT05411315
Title: Pragmatic Randomized Trial for Arterial Catheters in the Critical Care Environment
Acronym: GRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, David J. Feller-Kopman, Professor of Medicine, Geisel School of Medicine Chief, Pulmonary and Critical Care Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY02001496
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Mechanical Ventilation Complication; Arterial Thrombosis; Limb Ischemia; Shock; Hypotension; Bloodstream Infection; Vasopressor Adverse Reaction; Renal Failure
MeSH Terms: conditions — Shock; Hypotension; Sepsis; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restricted-use of arterial catheters (Experimental)
  Interventions: Other: Restricted-use of arterial catheter
- Standard-use of arterial catheters (Active Comparator)
  Interventions: Other: Standard-use of arterial catheter

INTERVENTIONS:
Other: Restricted-use of arterial catheter — The investigator will restrict the use of arterial catheters unless exclusion criteria is met.
  Arms: Restricted-use of arterial catheters
Other: Standard-use of arterial catheter — The investigator will allow standard-use of arterial catheters
  Arms: Standard-use of arterial catheters

SUMMARY:
Investigators will conduct a pragmatic randomized trial to investigate the non-inferiority of restricted use of invasive arterial lines compared to standard arterial line use.

DETAILED DESCRIPTION:
Patients in the medical intensive care unit (MICU) often receive arterial lines as standard of care, however there are little data to support this practice. Investigators will randomly assign consecutive weeks to either current practice(control) or to a more conservative practice of not placing invasive arterial lines except for limited indication indications as defined below (intervention). Patients entering during an intervention week will be treated according to the intervention practice throughout their ICU stay. Likewise, patients entering during a control week will be treated according to current standard practice.

Permuted block randomization will be used to assure equal numbers of intervention and control weeks. All outcome measures will be obtained through EPIC data analytics and post-hospitalization phone calls. Weekly randomization codes will be generated by the study statisticians and delivered to MICU staff via sealed envelopes to be opened at the beginning of each week.

ELIGIBILITY:
Inclusion Criteria:

* All subjects admitted to the medical intensive care unit

Exclusion Criterion:

* All subjects <18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Number of days hospitalized in the medical intensive care unit (length-of-stay) | inpatient hospitalization (approximately 1 to 30 days)
  Number of days hospitalized in the medical intensive care unit

SECONDARY OUTCOMES:
Number of days hospitalized in a non- medical intensive care unit (Hospital length-of-stay) | inpatient hospitalization (approximately 1 to 30 days)
  Number of days hospitalized in a non- medical intensive care unit
Number of days using a mechanical ventilator (Ventilator-days) | inpatient hospitalization (approximately 1 to 30 days)
  Number of days spent on a mechanical ventilator
Number of days using vasopressor medicines (vasopressor-days) | inpatient hospitalization (approximately 1 to 30 days)
  Number of days using vasopressor medicines
Number of blood transfusions received during hospitalization (packed red blood cell transfusions) | inpatient hospitalization (approximately 1 to 30 days) and receiving approximately 0 - 10 blood transfusions
  Number of blood transfusions received during hospitalization
Number of participants experiencing a bloodstream infection related to invasive arterial catheter use | inpatient hospitalization (approximately 1 to 30 days) and experiencing 0 to 1 bloodstream infections
  Number of participants experiencing a bloodstream infection related to invasive arterial catheter use
Number of participants experiencing a vascular injury related to the invasive arterial catheter | inpatient hospitalization (approximately 1 to 30 days)
  vascular injuries include hematoma formation, ischemic limb, false aneurysm, limb injury
Number of days subjects experiencing death within 28 days of medical intensive care unit while having received vasopressor medicines (28-day mortality while on vasopressors) | Inpatient or outpatient death within 1 to 28 days
  Number of days subjects experiencing death within 28 days of medical intensive care unit while having received vasopressor medicines
Number of days subjects experiencing death within 28 days of medical intensive care unit from any cause (28-day all-cause mortality) | Inpatient or outpatient death within 1 to 28 days
  Number of days subjects experiencing death within 28 days of medical intensive care unit from any cause
Number of days subjects experiencing death within 90 days of medical intensive care unit from any cause (90-day all-cause mortality) | Inpatient or outpatient death within 1 to 90 days
  The outcome of death that has occurred for subjects from all causes after 90 days
Number of patients experiencing renal failure while hospitalized | inpatient hospitalization (approximately 1 to 30 days)
  Renal failure is defined as any renal replacement therapy
Number of vasopressors used | Inpatient hospitalization (approximately 1 to 60 days)
  The quantity of vasopressors
Number of ABG measurements | Inpatient hospitalization (approximately 1 to 60 days)
  The total quantity of ABG labs sent

CONTACTS AND LOCATIONS:
Overall Officials: David Feller-Kopman, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No